CLINICAL TRIAL: NCT04342377
Title: Improving Preoperative Lung Cancer Staging Through the Canada Lymph Node Project: A Pan-Canadian Multicentered Crossover Trial
Brief Title: The Canada Lymph Node Score Project: A Crossover Trial
Acronym: CLNS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Health Sciences Centre, Winnipeg, Manitoba (Other); Royal Alexandra Hospital (Other); Toronto General Hospital (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Wael Hanna, Lead Investigator, McMaster University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: clns_10696
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Non-small Cell Lung Cancer Stage I; Non-small Cell Lung Cancer Stage II
Keywords: Mediastinal Staging; Nodal Disease; Endobronchial Ultrasound; Diagnostic Testing
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: A prospective pan-Canadian, multicentered, non-inferiority crossover study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective Targeted Sampling (Experimental): During patients' Endobronchial Ultrasound (EBUS) procedure, they will first undergo:
  Selective Targeted Sampling - endosonographic assessment of at least 3 mediastinal lymph node stations (4R, 4L, and 7) using the four criteria of the Canada Lymph Node Score (predictor of nodal disease during Endobronchial Ultrasound). Each lymph node will be assigned a CLNS ranging from 0 to 4. Triple Normal lymph nodes will be defined as those that appear normal on CT (diameter < 1 cm), AND normal on PET (SUV < 2.5), AND normal on EBUS (CLNS < 2). Lymph nodes that are found to be Triple Normal will be marked as "Not for Biopsy", whereas all other lymph nodes will be biopsied.
  Interventions: Diagnostic Test: Selective Targeted Sampling
- Systematic Sampling (Active Comparator): Upon completion of Systematic Targeted Sampling, all patients will crossover and receive the standard of care:
  Systematic Sampling - all lymph nodes previously marked as "Not for Biopsy" will be biopsied.
  At the conclusion of the EBUS procedure, all nodal stations would have been sampled as is mandated by current guidelines.
  Interventions: Diagnostic Test: Systematic Sampling

INTERVENTIONS:
Diagnostic Test: Selective Targeted Sampling — Mediastinal lymph nodes are assessed with the CLNS, and only those appearing malignant with the score are biopsied. Triple Normal lymph nodes (normal appearing on PET, CT and EBUS) are not biopsied.
  Other Names: STS
  Arms: Selective Targeted Sampling
Diagnostic Test: Systematic Sampling — All examined mediastinal lymph nodes are biopsied, regardless of whether they appear normal during PET, CT and EBUS.
  Other Names: SS
  Arms: Systematic Sampling

SUMMARY:
Before deciding on treatment for patients with lung cancer, a critical step in the investigation is finding out whether the lymph nodes in the chest contain cancer cells. This is accomplished with a biopsy of the lymph nodes through the airway wall, known as Endobronchial Ultrasound-guided Transbronchial Needle Aspiration. Guidelines require that every single lymph node in the chest be biopsied through a process called Systematic Sampling. However, emerging data suggests that the lymph nodes that appear benign on imaging and ultrasound do not need a biopsy. A proposed alternative to the inefficient Systematic Sampling is the simplified Selective Targeted Sampling of the lymph nodes, whereby only lymph nodes that look malignant are biopsied. This trial will evaluate the simplified Selective Targeted Sampling of lymph nodes and compare it to Systematic Sampling to see whether it is equally as effective in staging lung cancer.

DETAILED DESCRIPTION:
Treatment decisions in Non-Small Lung Cancer (NSCLC) are reliant on a thorough staging process that includes imaging with Computed Tomography (CT), Positron Emission Tomography (PET) and Systematic Sampling (SS) of mediastinal lymph nodes (LNs) by Endobronchial Ultrasound Transbronchial Needle Aspiration (EBUS-TBNA). Collectively, the results of these staging procedures dictate whether patients will be treated with surgery, radiation and/or chemotherapy. Current guidelines for SS through EBUS-TBNA mandate the biopsy of at least 3 mediastinal LN stations (4R, 4L and 7) in the chest, even if they appear normal on CT and PET scan. Despite improvements in diagnostic techniques and safety, LN biopsies remain onerous for the patient and costly to our healthcare system. SS is also unreliable, yielding inconclusive pathology results in 42.14% of cases, especially for Triple Normal LNs, which are LNs that appear normal on PET, and CT, and EBUS. In fact, SS results in mostly negative or inconclusive biopsies for Triple Normal LNs, which may be due in part to their very low probability (< 6%) of malignancy. As such, the researchers have proposed to replace the onerous and unreliable process of SS by a simpler Selective Targeted Sampling (STS) staging process. In STS, Triple Normal LNs will not be biopsied, due to the very high negative predictive value (NPV) of malignancy. STS follows the simple notion that only LNs that have the potential to be malignant should be biopsied, whereas LNs which are very likely benign (i.e. Triple Normal LNs) should not be biopsied.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both CT and PET scans completed prior to EBUS
* Suspected or confirmed NSCLC requiring mediastinal staging
* cN0-cN1 as indicated by CT and PET scans

Exclusion Criteria:

* Patients with cN0 disease AND peripheral tumors AND tumor < 2 cm in diameter, as they do not require mediastinal staging
* Evidence of cN2 disease or higher on CT and PET scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Non-Inferiority Margin between Selective Targeted Sampling and Systematic Sampling | 2 years
  A margin of 5% or less would be considered satisfactory for STS to be deemed non-inferior to SS.

SECONDARY OUTCOMES:
Diagnostic Statistics (between staging methods) | 2 years
  Sensitivity, specificity, negative predictive value and positive predictive value
Agreement (between staging methods) | 2 years
  Based on Cohen's Kappa statistics
Inconclusive Biopsy Rate | 2 years
  Percentage of lymph nodes with inconclusive pathology from biopsy
Diagnostic Yield (accuracy) | 2 years
  Proportion of lymph nodes with a pathological diagnosis for both sampling methods
Difference in Procedure Length | 2 years
  For each sampling method (in minutes)
Difference in Cost per Procedure | 2 years
  For each sampling method (sum of dollar costs for EBUS procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Waël C Hanna, MDCM, MBA, FRCSC, Principal Investigator — McMaster University
Locations (7):
- Canada (7):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Health Sciences Centre, Winnipeg, Manitoba
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CHUM Endoscopic Tracheo-bronchial and Oesophageal Center, Montreal, Quebec
  - MUHC Interventional Pulmonology Department, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No